CLINICAL TRIAL: NCT05303064
Title: A Phase 3, Randomized, Double-Blind, 52-Week Study of OLZ/SAM vs Olanzapine to Evaluate Weight Gain as Assessed by Change in BMI Z-Score in Pediatric Subjects With Schizophrenia or Bipolar I Disorder (ENLIGHTEN-Youth)
Brief Title: Study to Evaluate Weight Gain as Assessed by Change in BMI Z-score in Pediatric Subjects With Schizophrenia or Bipolar I Disorder
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Alkermes, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALKS 3831-A312
Record Dates: First submitted 2022-03-22; First posted 2022-03-31 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Schizophrenia; Bipolar I Disorder
Keywords: LYBALVI; Schizophrenia; Bipolar I Disorder; Pediatric; Olanzapine; Samidorphan
MeSH Terms: conditions — Schizophrenia | interventions — lybalvi; Olanzapine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 OLZ/SAM (Experimental): Fixed dose combination of olanzapine and samidorphan
  Interventions: Drug: OLZ/SAM
- Group 2 Olanzapine (Active Comparator): Fixed dose of olanzapine
  Interventions: Drug: Olanzapine

INTERVENTIONS:
Drug: OLZ/SAM — OLZ/SAM refers to the fixed dose combination of olanzapine and samidorphan. The starting dose of olanzapine will be 2.5 mg/day or 5 mg/day at the discretion of the Investigator with a maximum daily dose of 20mg/day. The starting dose of samidorphan will be 5 or 10 mg.
  Other Names: ALKS 3831, LYBALVI
  Arms: Group 1 OLZ/SAM
Drug: Olanzapine — The starting dose of olanzapine will be 2.5 mg/day or 5 mg/day at the discretion of the Investigator with a maximum daily dose of 20mg/day
  Arms: Group 2 Olanzapine

SUMMARY:
To compare changes in body mass index (BMI) Z-score following treatment with OLZ/SAM vs olanzapine

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 13 to 17 years with schizophrenia or aged 10 to 17 years with bipolar I disorder, diagnosed according to Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) criteria
* Subject is an outpatient or will be able to be treated on an outpatient basis (per Investigator judgement) by study Week 2
* Subject has reliable family/legal guardian support available for outpatient management
* Subject is either currently treated with olanzapine, or if treated with another antipsychotic, the subject has had an inadequate response (eg, unsatisfactory clinical response, AEs, or nonadherence to current medication) based on Investigator judgment
* Subject must not be a danger to self or others (per Investigator judgement)

Exclusion Criteria:

* Subject presents with a major depressive episode(bipolar I disorder) or other neuropsychiatric diagnosis (according to DSM-5 criteria) including schizoaffective disorder, current major depressive disorder that is untreated and/or unstable, or any other psychiatric condition that could interfere with participation in the study
* Subject has a history of seizure disorder (exception: history of febrile seizures), severe head trauma with loss of consciousness within the 12 months prior to Screening, or other clinically significant neurological condition within the 12 months prior to Screening
* Subject poses a current suicide risk as assessed by the Investigator or as confirmed by the baseline Columbia-Suicide Severity Rating Scale (C-SSRS)
* Subject has received olanzapine for >= 14 days during the month prior to screening, or has a history of poor or inadequate response to treatment with olanzapine
* Subject has taken opioid agonists within 14 days prior to Screening, or within 30 days prior to Screening (for long-acting opioid agonists)
* Subject anticipates needing to take opioid medication during the study period (eg, planned surgery, including oral surgery)
* Subject has taken opioid antagonists including naltrexone (any formulation) or naloxone within 60 days prior to Screening
* Subject has used a long-acting injectable antipsychotic medication within 3 injection cycles prior to Screening
* Subject has a BMI percentile >98th or <5th
* Subject has a diagnosis of diabetes mellitus or presents with prediabetes lab results at Screening (hemoglobin A1c [HbA1c] >= 6%)
* Subject has started a smoking cessation program within the 6 months prior to Screening or has joined a weight management program or has had significant changes in diet or exercise regimen within 6 weeks prior to Screening
* Subject has participated in a clinical study of an investigational product within the last 30 days prior to Screening

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 220 (Estimated)
Dates: Start 2022-06-30 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in body mass index (BMI) Zscore at week 12 | 12 weeks
  To compare changes in body mass index (BMI) Z-score following treatment with OLZ/SAM vs olanzapine

SECONDARY OUTCOMES:
Proportion of subjects with >=0.5 increase in BMI Z-score at Week 12 | 12 weeks
  To compare subjects with clinical significant BMI Z-score increase with OLZ/SAM vs olanzapine
Time to all-cause discontinuation of study drug over 52 weeks | Up to 52 weeks
  To compare time to all-cause discontinuation of study drug with OLZ/SAM vs olanzapine
Change from baseline in waist circumference | 12 weeks
  To compare the change from baseline in waist circumference with OLZ/SAM vs olanzapine
Change from baseline in Positive and Negative Syndrome Scale (PANSS) total score for patients with schizophrenia by visit | 12 weeks
  To compare the change from baseline in Positive and Negative Syndrome Scale (PANSS) total score with OLZ/SAM vs olanzapine for patients with schizophrenia
Change from baseline in Young Mania Rating Scale (YMRS) in patients with Bipolar I disorder | 12 weeks
  To compare the change from baseline in YMRS with OLZ/SAM vs olanzapine for patients with bipolar I disorder
Change from baseline in Children's Depression Rating Scale-Revised (CDRS-R) for patients with bipolar I disorder by visit | 12 weeks
  To compare the change from baseline in CDRS-R with OLZ/SAM vs olanzapine for patients with bipolar I disorder
Incidence of Adverse Events | Up to 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: David McDonnell, MD, Study Director — Alkermes, Inc.
Locations (43):
- United States (26):
  - Alkermes Investigator Site, Dothan, Alabama
  - Alkermes Investigator Site, Little Rock, Arkansas
  - Alkermes Investigator Site, Encino, California
  - Alkermes Investigator Site, Stanford, California
  - Alkermes Investigator Site, Upland, California
  - Alkermes Investigator Site, Colorado Springs, Colorado
  - Alkermes Investigator Site, Denver, Colorado
  - Alkermes Investigator Site, Hartford, Connecticut
  - Alkermes Investigator Site, Washington D.C., District of Columbia
  - Alkermes Investigator Site, Miami, Florida
  - Alkermes Investigator Site, Miami Lakes, Florida
  - Alkermes Investigator Site, Decatur, Georgia
  - Alkermes Investigator Site, Chicago, Illinois
  - Alkermes Investigator Site, Indianapolis, Indiana
  - Alkermes Investigator Site, Saint Charles, Missouri
  - Alkermes Investigator Site, Lincoln, Nebraska
  - Alkermes Investigator Site, Omaha, Nebraska
  - Alkermes Investigator Site, Paramus, New Jersey
  - Alkermes Investigator Site, New York, New York
  - Alkermes Investigational Site, Kinston, North Carolina
  - Alkermes Investigator Site, Cincinnati, Ohio
  - Alkermes Investigator Site, West Chester, Ohio
  - Alkermes Investigator Site, DeSoto, Texas
  - Alkermes Investigator Site, Fort Worth, Texas
  - Alkermes Investigational Site, Richmond, Virginia
  - Alkermes Investigator Site, Everett, Washington
- Argentina (4):
  - Alkermes Investigator Site, La Plata, Buenos Aires
  - Alkermes Investigator Site, Buenos Aires
  - Alkermes Investigator Site, Córdoba
  - Alkermes Investigator Site, Mendoza
- Brazil (5):
  - Alkermes Investigator Site, Fortaleza, Ceará
  - Alkermes Investigator Site, Curitiba, Paraná
  - Alkermes Investigator Site, Goiânia
  - Alkermes Investigator Site, Rio de Janeiro
  - Alkermes Investigator Site, São Paulo
- Colombia (4):
  - Alkermes Investigator Site, Barranquilla
  - Alkermes Investigator Site, Bello
  - Alkermes Investigator Site, Bogotá
  - Alkermes Investigator Site, Pereira
- Mexico (4):
  - Alkermes Investigator Site, Culiacán
  - Alkermes Investigator Site, Estado de México
  - Alkermes Investigator Site, León
  - Alkermes Investigator Site, Monterrey

IPD SHARING:
Plan to Share IPD: Undecided